CLINICAL TRIAL: NCT05416489
Title: Videolaryngoscopy Versus Direct Laryngoscopy for Positioning the Tracheal Tube During Percutaneous Tracheostomy: A Randomized Controlled Trial (VIDLARTRAQUEO).
Brief Title: C-MAC Videolaryngoscopy Versus Direct Laryngoscopy for Percutaneous Tracheostomy
Acronym: VIDLARTRAQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Manuel Taboada Muñiz, Clinical Professor, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIDLARTRAQUEO
Record Dates: First submitted 2022-02-24; First posted 2022-06-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Intubated Patients; Percutaneous Tracheostomy
Keywords: Tracheostomy; Critical care; Videolaryngoscopy; Direct laryngoscopy; Airway management

STUDY DESIGN:
Intervention Model Description: Randomized, controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional direct laryngoscopy technique (Active Comparator): Endotracheal tube will be removed before percutaneous tracheostomy using a traditional direct laryngoscopy technique.
  Interventions: Device: Laryngoscopy technique
- C-MAC videolaryngoscope technique (Active Comparator): Endotracheal tube will be removed before percutaneous tracheostomy using a C-MAC videolaryngoscope technique.
  Interventions: Device: C-MAC videolayngoscopy technique

INTERVENTIONS:
Device: C-MAC videolayngoscopy technique — Endotracheal tube will be removed before percutaneous tracheostomy using a C-MAC videolaryngoscopy.
  Arms: C-MAC videolaryngoscope technique
Device: Laryngoscopy technique — Endotracheal tube will be removed before percutaneous tracheostomy using a laryngoscopy
  Arms: Traditional direct laryngoscopy technique

SUMMARY:
When preparing an ICU patient for percutaneous dilational tracheostomy, correct positioning of the endotracheal tube is important. During the procedure, it is possible to puncture the cuff. Tracheal tube cuff puncture can lead to failure of ventilation, loss of positive end-expiratory pressure, and possible aspiration of gastric contents blood or secretions. To minimize the risk, in our ICU, we withdraw the endotracheal tube under direct laryngoscopic vision until the cuff is visible at the vocal cords. This maneuver would also facilitate insertion of the Seldinger needle and insertion of the tracheostomy tube below the endotracheal tube. However, this maneuver to remove the endotracheal tube under direct laryngoscopy can sometimes be difficult. ICU patients present frecuently difficult laryngoscopic vision due to airway edema or secretions. In ICU, the videolaryngopy has been shown to be superior to direct laryngoscopy in visualization the upper airway, allowing better laryngoscopic vision.

DETAILED DESCRIPTION:
The investigators aim to compare C-MAC videolaryngoscopy versus conventional direct laryngoscopy for positioning the tracheal tube to facilitate insertion of the Seldinger needle and the tracheostomy tube below the endotracheal tube during percutaneous tracheostomy.

ELIGIBILITY:
Inclusion Criteria:

* ICU intubated patients that require a percutaneous dilational tracheostomy for clinical reasons (prolonged mechanical ventilation, airway protection or weaning failure).

Exclusion Criteria:

* Patients younger than 18 years and older than 85 years
* Trachea and neck abnormalities.
* Soft tissue infection in the neck.
* History of neck surgery.
* Coagulation disorders or changes in coagulation parameters (platelet count < 50.000 mm3, an activated partial thromboplastin time 1.5-fold longer than the control value, and international normalized ratio > 1.5).
* Consent refusal for participating in the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Introduction of the Seldinger needle below the endotracheal tube | during the procedure
  Percentage of patients in whom the introduction of the Seldinger needle is below the tip of the endotracheal tube

SECONDARY OUTCOMES:
Puncture of the cuff of the endotracheal tube with the Seldinger needle | during the procedure
  Percentage of patients suffering puncture the cuff of the endotracheal tube with the Seldinger needle
patients who need to remove the endotracheal tube to introduce the percutaneous tracheostomy cannula | during the procedure
  Percentage of patients who need to remove the endotracheal tube to introduce the percutaneous tracheostomy cannula
Laryngoscopy vision using de Modified Cormack-Lehane grade of glottic view | during the procedure
  Differences in laryngoscopy vision using de modified Cormack-Lehane grade of glottic view
  Modified Cormack-Lehane grade of glottic view:
  I: full view of the glottis (better outcome) IIa: partial view of the glottis IIb: arytenoid or posterior part of the vocal cords just visible III: only epiglottis visible IV: neither glottis nor epiglottis visible (worse outcome)
Difficulty of removing the endotracheal tube | during the procedure
  Differences in the difficulty of removing the endotracheal tube due to poor visualization, secretions....
  Operator-assessed subjective difficulty of removing the endotracheal tube: No difficulty, mild difficulty, moderate difficulty, severe difficulty.
Difficulty of performing percutaneous tracheotomy | during the procedure
  Differences in the difficulty of performing percutaneous tracheotomy Operator-assessed subjective difficulty of performing percutaneous tracheotomy: No difficulty, mild difficulty, moderate difficulty, severe difficulty.
Complications | during the ICU stay
  Percentage of complications

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Hospital of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson-Obaseki S, Veljkovic A, Javidnia H. Complication rates of open surgical versus percutaneous tracheostomy in critically ill patients. Laryngoscope. 2016 Nov;126(11):2459-2467. doi: 10.1002/lary.26019. Epub 2016 Apr 14. PMID 27075530